CLINICAL TRIAL: NCT06704009
Title: A Randomized, Open-Label, Parallel-group, Multicenter Phase 1/2 Study to Evaluate the Safety and Exploratory Efficacy of NT-101 Topical Ophthalmic Solution in Patients With Wet Age-Related Macular Degeneration (AMD)
Brief Title: NT-101 Topical Ophthalmic Solution in Patients With Wet AMD
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NexThera Co., Ltd. (Industry)
Collaborators: KCRN Research, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NT101-AMD-001
Record Dates: First submitted 2024-11-18; First posted 2024-11-25 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Wet Age Related Macular Degeneration; Wet AMD
Keywords: wet AMD; Age related Macular Degeneration; Eyedrop
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NT-101 Low Dose (Experimental)
  Interventions: Drug: NT-101 Low Dose
- NT-101 High Dose (Experimental)
  Interventions: Drug: NT-101 High Dose

INTERVENTIONS:
Drug: NT-101 Low Dose — Low concentration of NT-101 (0.05 mM)
  Arms: NT-101 Low Dose
Drug: NT-101 High Dose — High concentration of NT-101 (0.2 mM)
  Arms: NT-101 High Dose

SUMMARY:
Phase 1/2 Trial NT-101 Topical Ophthalmic Solution in Patients with Wet Age-Related Macular Degeneration (AMD)

ELIGIBILITY:
Inclusion Criteria:

1. Subject who is male or female ≥ 50 years of age at Screening.
2. Choroidal neovascularization (CNV) lesions secondary to AMD that affected the central subfield in the study eye that meets the following criteria at Screening:

   * Total area of CNV (including both classical and occult) comprising > 50% of the total lesion area on FA
   * Leakage covering > 50% of the total lesion area on FA
   * Intraretinal and/or subretinal fluid affecting the central subfield visible on OCT.

   If fluid is not visible due to previous treatment, earlier documented OCT images showing fluid for diagnosing wet AMD can be reviewed to fulfill this criterion.

   • No atrophy or fibrosis involving the center of the fovea.
3. BCVA between 25 and 78 letters, inclusive, in the study eye at Screening using ETDRS testing, with BCVA decrement primarily attributable to wet AMD.
4. Either no previous treatment in the study eye with anti-VEGF therapy (treatment naïve) or previously treated study eye with adequate washout from the baseline visit as defined below:

   * Lucentis (ranibizumab): 30-day washout
   * Avastin (bevacizumab): 30-day washout
   * Eylea (aflibercept): 60-day washout
   * Eylea (aflibercept) high dose 8mg: 90-day washout
   * Vabysmo (faricimab-svoa): 90-day washout
   * Biosimilars

     * Byooviz (ranibizumab-nuna): 30-day washout
     * Cimerli (ranibizumab-eqrn): 30-day washout
5. Demonstrate the ability to instill eye drops (by the subject or caregiver) in the study eye, express willingness to comply with the dosing regimen, and commit to attending all study visits.
6. Understands and voluntarily signs an informed consent form.
7. Female participants of childbearing potential and male participants able to father children must have (or have a partner who has) had a hysterectomy or vasectomy, be completely abstinent from intercourse, or agree to practice two acceptable methods of contraception throughout the course of the study and 3 months after their last study administration. Acceptable methods of contraception include :

   * hormonal contraception (i.e., birth control pills, injected hormones, dermal patch, or vaginal ring),
   * intrauterine device,
   * barrier methods (diaphragm, condom) with spermicide, or
   * surgical sterilization (hysterectomy or tubal ligation).

Exclusion Criteria:

1. Subject who has the following illness or abnormal laboratory test values at

   Screening:
   * Uncontrolled hypertension (systolic > 180 mmHg or diastolic > 100 mmHg) despite optimal medical regimen
   * Uncontrolled diabetes (HbA1c > 12.0%)
   * Total bilirubin > 1.5 × Upper Limit of Normal (ULN)
   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 x ULN
   * Prothrombin time (PT) > 1.5 x ULN
   * Hemoglobin (Hb) < 10 g/dL (male); Hb < 9 g/dL (female)
   * Platelets < 100 x 103/μL
   * Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m2
   * Positive results for Human Immunodeficiency Virus (HIV) or Hepatitis B or C viruses
2. Other clinically significant abnormal lab values per Investigator's judgement.
3. Subject who has a medical condition that, in the opinion of the Investigator, would preclude participation in the study (e.g., unstable medical status including psychiatric disorder, cardiovascular disease, poor glycemic control, and significant medical condition including end-stage renal disease and severe liver diseases).
4. History of stroke or myocardial infarction within 6 months prior to Screening.
5. Subject who has had major surgery within 3 months prior to Screening.
6. Pregnant or breastfeeding or intended to become pregnant during the study.
7. Subject with known hypersensitivity to any active substance or excipients of the investigational product, fluorescein, dilating eye drops, or any of the anesthetic and antimicrobial drops.
8. Treatment with investigational therapy or participation in any other type of interventional trial within 30 days before Screening.
9. Subject who has a history of AMD treatment in the study eye with Beovu® (brolucizumab) or photodynamic therapy.
10. CNV in the study eye secondary to other causes or subject who has an ocular condition (other than AMD) that, in the opinion of the Investigator, may limit visual acuity improvement during the course of the study (e.g., ocular histoplasmosis, trauma, pathological myopia, angioid streaks, choroidal rupture, multifocal choroiditis, congenital eye malformations, retinal pigment epithelial tear, or posterior uveitis etc.)
11. Media opacities or abnormalities in the study eye that would preclude visualization of the retina.
12. Subject who has a history of retinal detachment or retinal detachment repair surgery in the study eye.
13. Subject who has a history of yttrium aluminum garnet (YAG) capsulotomy performed within 2 months prior to randomization in the study eye.
14. Uncontrolled glaucoma in either eye (IOP > 25 mmHg despite treatment with a standard regimen of antiglaucoma medications), with exceptions allowed at the Investigator's discretion.
15. Any active intraocular or periocular infection or active intraocular inflammation (e.g., infectious conjunctivitis, keratitis, scleritis, endophthalmitis, infectious blepharitis, uveitis) in either eye on Screening.
16. Subject who has a history of vitrectomy in the study eye.
17. Subject who has a history of ocular surgery in the study eye (including cataract extraction, any intraocular surgery, etc.) within 3 months prior to Screening or anticipated within the next 6 months following randomization.
18. Subject who has any history of intraocular inflammation in either eye other than what would be expected in the normal post-operative course following prior routine ocular surgery such as cataract surgery.
19. Subject who has other retinal pathologies in the study eye that would interfere with vision, such as evidence of diabetic macular edema or diabetic retinopathy (defined as more than one microaneurysm).
20. Non-study eye with a BCVA worse than 20 letters at Screening using ETDRS testing.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Number and Severity of Treatment-Emergent Adverse Events (TEAEs) up to Week 8 | 8 weeks

SECONDARY OUTCOMES:
Change in CST in the Study Eye | Week 4 compared to baseline
  Measured by: SD-OCT | Unit: Micrometers (µm)
Change in ETDRS BCVA Letter Score in the Study Eye | Week 4 compared to baseline
  Unit: Letter Score
Change in IOP in the Study Eye | Week 4 compared to baseline
  Unit: Millimeters of Mercury (mmHg)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Elman Retina Group, Rosedale, Maryland
  - Duke Eye Center, Durham, North Carolina
  - Erie Retina Research, Erie, Pennsylvania
  - Texas Retina Associates, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No